CLINICAL TRIAL: NCT03232437
Title: A Multicenter Study to Evaluate the External Precision of the Aina HbA1c Monitoring System in Quantitative Measurement of Glycosylated Hemoglobin (HbA1c)
Brief Title: Reproducibility of HbA1c Measurement on the Aina HbA1c Monitoring System
Status: Completed | Type: Observational
Sponsor: Jana Care (Industry)
Collaborators: The Forsyth Institute (Other); Orange County Research Center (Other); ActivMed Practices & Research (Other)
Responsible Party: Sponsor
Other Study IDs: A1C-FI-001; A1C-OCRC-001 (Other: JanaCare); A1C-AM-001 (Other: JanaCare)
Record Dates: First submitted 2017-07-12; First posted 2017-07-28 (Actual); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Diabetes
Keywords: HbA1c
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood collected in EDTA vacutainers, aliquoted into smaller vials for shipment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Aina HbA1c Monitoring System — Monitoring test for quantitative determination of HbA1c

SUMMARY:
A three site study to evaluate the reproducibility of the Aina HbA1c Monitoring System in quantitative determination of glycosylated hemoglobin (HbA1c) took place at the following sites:

1. Forsyth Institute in Cambridge, MA
2. Orange County Research Center in Tustin, CA
3. ActivMed Practices & Research in Methuen, MA

DETAILED DESCRIPTION:
Each site tested three identical samples of HbA1c, at three different levels of HbA1c measurement. Samples were drawn at the Forsyth Institute, received and blinded by the Sponsor, and returned to Forsyth Institute for testing. Samples were tested in triplicate, twice per day, over the course of five days, by three trained operators.

ELIGIBILITY:
Inclusion Criteria:

* Agree to the terms of this consent form
* Sign this consent form
* Be 18 years or older
* Have an HbA1c measured by a reference method within the last three months or based on medical history that is expected to fall in the range of 4 to 15%
* Provide blood samples from your arm and finger
* Come in in the morning of the study visit

Exclusion Criteria:

* Not have a recent history of anemia or hemoglobin concentration above 20%
* Not be pregnant
* Not have previously given a blood sample to the Study Sponsor for a study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy and Diabetic patients
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2017-06-21 (Actual); Study Completion 2017-06-21 (Actual)

PRIMARY OUTCOMES:
Precision (as measured by %CV) of HbA1c measurements | Each sample was measured in triplicate, twice per day, over the course of five days
  HbA1c measured on 3 samples on the Aina HbA1c Monitoring System by 3 operators at each site.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Hasturk, PhD, Principal Investigator — Forsyth Institute; Joel Neutel, MD, Principal Investigator — Orange County Research Center; Michael McCartney, MD, Principal Investigator — ActivMed Practices & Research
Locations (3):
- United States (3):
  - Orange County Research Center, Tustin, California
  - The Forsyth Institute, Cambridge, Massachusetts
  - ActivMed Practices & Research, Methuen, Massachusetts

IPD SHARING:
Plan to Share IPD: No